CLINICAL TRIAL: NCT05346731
Title: Efficacy and Safety Addition of Low Dose Olanzapine to the Standard Prophylaxis of Nausea and Vomiting Induced by Highly-emetogenic Chemotherapy in Children and Adolescents (OZONE-V)
Brief Title: Low Dose Olanzapine to the Prophylaxis of Nausea and Vomiting Induced by Chemotherapy in Children and Adolescents
Acronym: OZONE-V
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OZONE-V
Record Dates: First submitted 2022-04-14; First posted 2022-04-26 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Ondansetron; Dexamethasone; Aprepitant; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): 1. Weight category 30-40 kg will receive: dexamethasone (5 mg/m2), ondansetron (0.15 mg/kg), aprepitant (80 mg)
  2. Weight category > 40 kg will receive:
  dexamethasone (5 mg/m2), ondansetron (0.15 mg/kg), aprepitant (125 mg) Note: aprepitant at a dose of 80 mg/day. applied for another 2 days, regardless of the number of days of chemotherapy.
  Interventions: Drug: Ondansetron; Drug: Dexamethasone; Drug: Aprepitant
- Olanzapine (Experimental): 1. Weight category 30-40 kg will receive:
     dexamethasone (5 mg/m2), ondansetron (0.15 mg/kg), aprepitant (80 mg), olanzapine (2.5 mg)
  2. Weight category > 40 kg will receive: dexamethasone (5 mg/m2), ondansetron (0.15 mg/kg), aprepitant (125 mg), olanzapine (2.5 mg for <55 kg, 5 mg for >55 kg) Note: aprepitant at a dose of 80 mg/day. applied for another 2 days, regardless of the number of days of chemotherapy.
  Interventions: Drug: Ondansetron; Drug: Dexamethasone; Drug: Aprepitant; Drug: Olanzapine

INTERVENTIONS:
Drug: Ondansetron — Ondnsetron will be administered at a dose of 0.15 mg/kg IV/PO every 8 hours on the day(s) of chemotherapy and 3 days after completion of chemotherapy
Drug: Dexamethasone — Dexamethasone will be administered at a dose of 5 mg/m2 intravenously/orally once on the day(s) of chemotherapy and 3 days after completion of chemotherapy;
Drug: Aprepitant — Aprepitant will be administered based on body weight:
  body weight 30-40 kg: days 1-3 - 80 mg orally; body weight > 40 kg: day 1 - 125 mg orally, days 2, 3 - 80 mg orally
Drug: Olanzapine — Olanzapine will be administered at a dose of 0.07 mg/kg orally on the day(s) of chemotherapy and 3 days after completion of chemotherapy (rounded up to the maximum multiple of 2.5 mg, maximum daily dose of 5 mg).
  Arms: Olanzapine

SUMMARY:
Chemotherapy-induced nausea and vomiting continues to be a significant problem in children and adolescents. Standard antiemetic therapy, including a 5-HT3 antagonist, aprepitant, and a corticosteroid, achieves complete control in less than 50% of patients. Studies have shown that the addition of large doses of olanzapine improves control, including in children and adolescents. However, olanzapine has not yet been included in standard recommendations in the pediatric population. Studies in adults indicate that the dose of the drug can be halved without loss of effectiveness and with a decrease in toxicity. This open-label, randomized, phase III trial evaluates the efficacy and safety of adding low-dose olanzapine to standard prevention of nausea and vomiting induced by highly emetogenic chemotherapy in children and adolescents.

DETAILED DESCRIPTION:
After signing informed consent, eligible patients are randomized with stratification (previously received or not received high emetogenic therapy; regimens with and without cisplatin) to receive the first cycle of highly emetogenic chemotherapy with standard prophylaxis (5-HT3 receptor antagonist, dexamethasone, aprepitant) with or without addition of 0.07 mg/kg olanzapine (rounded to multiples of 2.5 mg, maximum 5 mg). During chemotherapy and 120 hours after its completion, patients are assessed for the presence and absence, as well as the severity of CINV, the need for "rescue" therapy, and the development of adverse events. In the future, patients undergo a similar course of highly emetogenic chemotherapy with a change in the antiemetic prophylaxis option - crossover (patients who received an olanzapine regimen as antiemetic prophylaxis after the first cycle of chemotherapy receive treatment without it, patients who received prophylaxis without olanzapine receive a second cycle of therapy with olanzapine). After this cycle, the presence and absence, as well as the severity of CINV, the need for salvage therapy, the development of adverse events are assessed and, additionally, at the end of the cycle, patients are asked about the preferred option for further antiemetic prophylaxis (the regimen with olanzapine, no olanzapine, or no preferences).

ELIGIBILITY:
Inclusion Criteria:

1. Age from 5 to 18 years.
2. Body weight ≥ 30 kg.
3. Confirmed diagnosis of malignancy.
4. Planned at least 2 cycles of highly emetogenic chemotherapy according to the Pediatric Ontario Cancer Group (POGO) emetogenicity classification.
5. ECOG status < 3.
6. Adequate function of internal organs (bilirubin < 1.5 upper limit of normal (ULN), ALT and AST <2.5 ULN, creatinine < 1.5 ULN).
7. Ability to swallow study drug.
8. The presence of a written voluntary informed consent of the patient and / or his legal representative.

Exclusion Criteria:

1. Treatment with olanzapine or another antipsychotic drug within the last 30 days.
2. Planned use of antibiotics from the group of fluoroquinolones or other drugs that have drug interactions with olanzapine and other drugs used in the study (amifostin, citalopram, CYP1A2 inducers or inhibitors).
3. The presence of intensive CINV against the background of a previous similar cycle of chemotherapy, which does not allow prescribing standard antiemetic prophylaxis upon inclusion in the study.
4. The presence of a convulsive syndrome.
5. Hypersensitivity to olanzapine or other drugs used in the study.
6. Uncontrolled arterial hypertension or cardiovascular disorders, uncontrolled diabetes mellitus, or other diseases and conditions that, in the opinion of the physician, preclude study therapy.
7. The presence of other factors (other than ongoing highly emetogenic therapy) that can cause the development of CINV (radiotherapy to the abdominal cavity or pelvis 1 week or less before inclusion in the study, obstruction of the gastrointestinal tract, uncontrolled intracranial hypertension, etc.).
8. Severe CINV of any intensity 24 hours or less before the first dose of chemotherapy.
9. Pregnancy or breastfeeding.
10. Planned use of systemic glucocorticosteroids at the time of inclusion in the study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Complete control of vomiting | up to 21 days
  proportion of patients who did not have episodes of vomiting and/or use of additional antiemetic drugs (rescue therapy) during the chemotherapy cycle and within 120 hours after its completion
Patient preference | up to 42 days
  Proportion of patients who, after crossover, chose to continue treatment with an experimental regimen including olanzapine
Adverce events | up to 42 days
  Percentage of patients with grade 3-4 adverse events according to CTCAE v. 5.0. [Time frame: day(s) of chemotherapy administration and 120 hours after chemotherapy administration]

SECONDARY OUTCOMES:
Complete control of acute vomiting | up to 21 days
  Proportion of patients who did not have episodes of vomiting and/or use of additional antiemetic drugs (rescue therapy) during the chemotherapy cycle and within 24 hours after its completion
Complete control of chemotherapy-induced nausea and vomiting (CINV) | up to 21 days
  Proportion of patients who did not experience nausea (PeNAT score 1) and/or vomiting and/or use of additional antiemetics (rescue therapy) during the chemotherapy cycle and within 120 hours after its completion

CONTACTS AND LOCATIONS:
Locations (1):
- Zhukov Nikolay, Moscow, Russia